CLINICAL TRIAL: NCT05141240
Title: A Real-world Analysis of Concomitant Medication Use Among Metastatic Breast Cancer Patients Treated With CDK4/6 Inhibitors
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AUS64
Record Dates: First submitted 2021-11-11; First posted 2021-12-02 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Concomitant medication,; drug-drug interaction,; CDK4/6 inihibitor,; HR+/HER2-metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ribociclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Ribiciclib
- Palbociclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Palbociclib
- Abemaciclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Ribiciclib — Participants who initiated CDK4/6i therapy
  Groups: Ribociclib
Drug: Palbociclib — Participants who initiated CDK4/6i therapy
  Groups: Palbociclib
Drug: Abemaciclib — Participants who initiated CDK4/6i therapy
  Groups: Abemaciclib

SUMMARY:
This is a retrospective cohort study to assess the real-world analysis of concomitant medication use among metastatic breast cancer patients treated with CDK4/6 inhibitors utilizing the US Optum research administrative claims database.

DETAILED DESCRIPTION:
This is a retrospective cohort study utilizing the US Optum research administrative claims database. Adult female patients who had HR+/HER2- mBC were identified and included in the study. These patients were stratified into three cohorts based on the first CDK4/6i received (ribociclib, palbociclib, or abemaciclib).

* Study period: Period during which all relevant medical and pharmacy information in the database was retrieved
* Index event identification period: time frame during which index treatment was identified
* First CDK4/6i: the date on which patients initiated their first treatment after being diagnosed with HR+/HER2- mBC; this date was considered as the index date
* Baseline period: Time frame during which patient characteristics, prior mBC treatments, and concomitant treatments received by CDK4/6i-naïve patients were evaluated
* Follow-up period: time frame on and after the index date during which patients' treatments and dosing patterns were observed

Establishment of baseline period Health plan enrollment in the three months prior to the index treatment was included in the baseline period. Patient demographics, clinical characteristics, National Cancer Institute (NCI) comorbidity index, concomitant medication use that can potentially lead to a DDI, and other BC treatments prior to the index treatment were evaluated during this period.

Establishment of follow-up period Patients were observed for ≥3 months starting from the index date until the end of the study period or continuous enrollment or until the time when patients switched to another therapy (including another CDK4/6i), whichever came first. Dosing patterns for CDK4/6i were evaluated in the follow-up period. Analyses were conducted at key time points of 3, 6, and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Treated with CDK4/6i from 2015-02-01 to 2019-06-30
* ≥2 claims with a BC diagnosis recorded ≥30 days apart from the index date
* ≥2 claims with an mBC diagnosis, with a time interval between the first BC diagnosis date and the first mBC diagnosis date no longer than 30 days
* Female patients aged ≥18 years
* Continuous health plan enrollment for ≥3 months prior to the index date and ≥3 months post-index date

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women with HR+/HER2- mBC
Study Population: Study analyses were conducted among adult women with HR+/HER2- mBC receiving ribociclib, palbociclib, or abemaciclib, regardless of the line of therapy. Patients were identified from the US Optum Claims Data.
Sampling Method: Probability Sample
Enrollment: 4650 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with a prescription fill of ribociclib, palbociclib, or abemaciclib | Index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time)
  Distribution of patients with a prescription fill of ribociclib, palbociclib, or abemaciclib at index treatment date will be present by frequency among all patients treated with CDK4/6
Number of participants who took concomitant medications in baseline period, by drug name | Baseline period (3 months)
  Number of patients taking a concomitant medication/s during baseline period that can potentially lead to a drug-drug interactions (DDI) with a CDK4/6 inhibitor use with each CDK4/6 inhibitor in the follow-up period.
Number of participants who took concomitant medications in follow-up period, by drug name | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Number of patients taking a concomitant medication/s during baseline period that can potentially lead to a drug-drug interactions (DDI) with a CDK4/6 inhibitor use with each CDK4/6 inhibitor in the follow-up period.
Number of participants with no use of concomitant medications | Baseline period (3 months)
  Adherence to concomitant medications during the baseline period was reported
Number of participants with proportion of days covered (PDC) >80% | Baseline period (3 months)
  Adherence to concomitant medication during the baseline period will be assessed using the proportion of days covered (PDC):
  PDC = total days of filled or refilled concomitant Rx in baseline period / total number of days in baseline period
Number of participants with proportion of days covered (PDC) ≤80% | Baseline period (3 months)
  Adherence to concomitant medication during the baseline period will be assessed using the proportion of days covered (PDC):
  PDC = total days of filled or refilled concomitant Rx in baseline period / total number of days in baseline period
Number of other breast cancer medications used | Baseline period (3 months)
  Number of other breast cancer medications used in baseline period, by drug class (HR+/Endocrine, Chemotherapy, Other treatments), for breast cancer regimens was reported

SECONDARY OUTCOMES:
Mean starting dose for each CDK4/6 | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Distribution of starting dose and mean starting dose for each CDK4/6 was reported to describe dosing and treatment patterns associated with ribociclib, palbociclib, and abemaciclib patients
Number of participants who had any dose change (increase, decrease) | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Number of patients with change in dose by each CDK4/6 inhibitor (ribociclib, palbociclib, and abemaciclib) in the follow-up period was reported
Number of participants who had a dose increase | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Number of patients with change in dose by each CDK4/6 inhibitor (ribociclib, palbociclib, and abemaciclib) in the follow-up period was reported
Number of participants who had a dose decrease | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Number of patients with change in dose by each CDK4/6 inhibitor (ribociclib, palbociclib, and abemaciclib) in the follow-up period was reported
Number of participants discontinuing each CDK4/6i (ribociclib, palbociclib, or abemaciclib) | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Rate of discontinuation of ribociclib, palbociclib, or abemaciclib in the follow-up period was reported
Median duration of treatment (in months) by each CDK4/6i (ribociclib, palbociclib, or abemaciclib) | From index date (defined as the prescription fill for ribociclib, palbociclib, or abemaciclib for the first time) to the end of follow-up period (12 months post index date)
  Duration of treatment with ribociclib, palbociclib, or abemaciclib, defined as discontinuation of each index CDK 4/6 treatment during the follow-up period was reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CLEE011AUS64 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17880